CLINICAL TRIAL: NCT05410106
Title: A Single Centre, Open-label, Feasibility Randomised Controlled Trial to Evaluate Gastric Microaspiration in Critically Ill Patients Intubated Using the Venner PneuX System Compared to Standard of Care Using Pepsin Biomarker (VAP-X)
Brief Title: Ventilator Aspiration With PneuX (PneuX vs Standard Care Feasibility RCT)
Acronym: VAP-X
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21/NOV/8290
Record Dates: First submitted 2022-05-18; First posted 2022-06-08 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-08

CONDITIONS: Ventilator Associated Pneumonia; Aspiration; Infections; Ventilator Lung
Keywords: Ventilator Associated Pneumonia; endotracheal tube; Aspiration
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections

STUDY DESIGN:
Intervention Model Description: Feasibility, 2-arm, parallel, randomised controlled trial
Who Masked: Participant
Masking Description: Due to the nature of the interventional device it is not possible to blind the care providers or outcome assessors to the intervention group. The trial participants will be unconscious/sedated for the duration of the period that the PneuX device or standard ETT is in place and therefore will be unaware of their allocation. Samples sent to the laboratory for analysis will be anonymised using individual deidentified numbers for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PneuX endotracheal tube (Experimental): Patients will be intubated using the PneuX endotracheal tube system
  Interventions: Device: PneuX Endotracheal Tube
- Standard care (Active Comparator): Patients will be intubated using standard endotracheal tube (Taperguard, Covidien).
  Interventions: Device: Standard care (Taperguard, Covidien)

INTERVENTIONS:
Device: PneuX Endotracheal Tube — The PneuX Endotracheal Tube is a CE marked device produced by Venner. The purpose of this product is to provide invasive ventilation for patients in the ICU. The defining features of the intervention treatment are the multi-modal approach to prevent microaspiration during long term ventilation.
  Other Names: Venner PneuX System
  Arms: PneuX endotracheal tube
Device: Standard care (Taperguard, Covidien) — Standard care is to intubate patient using the Taperguard endotracheal tube (ETT). The Taperguard ETT is designed with a tracheal shaped cuff made of PVC. This has a single lumen subglottic port.
  Arms: Standard care

SUMMARY:
This is a single centre, open-label, feasibility randomised controlled trial. The study aims to assess the feasibility of conducting an RCT to compare the PneuX ETT with standard care in hospitalised patients requiring mechanical ventilation. The patient population for this study are those who are experiencing critical illness requiring intubation and ventilatory support. Patients will be randomised in equal proportions into one of 2 arms: to be intubated using a Venner PneuX Endotracheal Tube (ETT) or using the standard tube. For this feasibility study, a total of 50 patients will be randomised into two groups (25 in each). All patients will be recruited at a single site (University Hospital of Wales, part of Cardiff & Vale UHB). The study will investigate several feasibility measures including recruitment, delivery of the intervention (including device-related adverse events), acceptability and adherence to the intervention and sampling, use of Peptest to measure microaspiration events, rate of pepsin positive samples, rate of tracheobronchial colonisation, volume of sub-glottic aspirate, rate of VAP, length of ICU and hospital stay, demonstrate the validity of study documentation and provide preliminary data for 50 patients. The data will inform the pilot and main phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old (no upper age)
* Patient required endotracheal intubation
* Expect to remain intubated for 24 hours post randomisation

Exclusion Criteria:

* The person intubating the patient assesses that the patient has already aspirated.
* GCS 7 or less on presentation to hospital
* Patient is pregnant
* Patient has tracheostomy
* Patient has gastrectomy
* Patients who have been intubated prior to arrival at hospital
* Patients who are already endotracheally intubated and require a tube change.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess if a recruitment rate of 50 patient annually is achievable and identify any barriers to recruitment | Through study completion, an average of 1 year
  The recruitment rate will be assessed using the "screening and recruitment log" which will record the number of patients recruited each month and reasons for non-recruitment will be described

SECONDARY OUTCOMES:
To assess the feasibility of delivering the study intervention | Duration of study treatment (typically 4-7 days)
  Any issues experienced when using the study device at any point during the study will be recorded in the CRF, including device-related complications.
Number of participants with a failed pepsin test | Duration of study treatment (typically 4-7 days)
  Any issues such as failed sampling or failed testing will be recorded in case report form
Number of participants with a positive pepsin tracheal aspirate sample using Peptest | Duration of study treatment (typically 4-7 days)
  The proportion of tracheal aspirate samples which are positive for the presence of pepsin using the Peptest test
Volume of sub-glottic aspirates | Duration of study treatment (typically 4-7 days)
  The volume of the sub-glottic aspirates will be measured every 24 hours
Rate of tracheobronchial colonization | Duration of study treatment (typically 4-7 days)
  Tracheobronchial colonization (no. colony forming units/ml) present in sputum samples will be measured by culture on days 3 and 7
Proportion of patients who require antibiotics | 28 days
  The following will be assessed: antibiotic prescribed, indication for use, number of days administered
Rate of Ventilator Associated Pneumonia (VAP) | 28 days
  Number of patients with VAP diagnosis. Clinical Pulmonary Infection Score (CPIS) used to predict VAP. CPIS >6 will be used to define confirmation of VAP. Measured daily after 48 hours of intubation
Time spent on the ventilator | Duration of study treatment (typically 4-7 days)
  Days spent with mechanical ventilation in ICU (from time/date of intubation to time/date of extubation or 28 days)
Number of days spent in ICU and hospital | 28 days
  Length of stay in ICU and length of stay in hospital measured in days from ventilation
Rate of in-hospital mortality | 28 days
  Number of patients who die in hospital up to 28 days after entry into ICU
Rate of compliance with measuring and documenting cuff pressure | Duration of study treatment (typically 4-7 days)
  Documentation of cuff pressures in both arms of study. Cuff pressure in standard care will be measured every 12 hours. Assessment of intervention arm will have documentation that pressure has been maintained hourly either via the continual cuff pressure monitor or manually.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wise, Study Chair — Cardiff and Vale University Health Board; Matthew Wise, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No